CLINICAL TRIAL: NCT00491946
Title: A Pharmacokinetic Study of Actinomycin-D and Vincristine in Children With Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPRU 10762
Record Dates: First submitted 2007-06-22; First posted 2007-06-26 (Estimated); Last update posted 2007-06-26 (Estimated); Status verified 2007-06

CONDITIONS: Cancer
Keywords: Cancer; Actinomycin; Vincristine
MeSH Terms: conditions — Neoplasms | interventions — Dactinomycin; Vincristine

INTERVENTIONS:
Drug: Actinomycin-D
Drug: Vincristine

SUMMARY:
To obtain a preliminary characterization of the plasma PK and metabolites of actinomycin-D in children with cancer.

DETAILED DESCRIPTION:
There is a fundamental lack of knowledge regarding optimal dosing of anti-cancer agents for young children with cancer, with resultant increased risk of morbidity, mortality and inferior outcome. Of the anti-cancer agents used frequently in infants and young children, the drug with the least amount of knowledge is actinomycin-D. Actinomycin-D, has been used for the treatment of several childhood cancers since the 1960s. Despite its longstanding and widespread use in pediatric oncology, there is virtually no pharmacokinetic information from which safe and appropriate age-based pediatric dosing can be derived. Actinomycin-D is an integral component of rhabdomyosarcoma and Wilms tumor therapy, and pediatric oncologists will continue to administer the durg despite the gap in knowledge.

ELIGIBILITY:
Inclusion Criteria:

* 6 months - 18 years
* Due to receive actinomycin-D as a component of cancer treatment
* Central venous catheter (e.g. Port-a Cath, Broviac)
* Informed consent of parent or legal guardian and patient assent when appropriate

Exclusion Criteria:

* Serious illness other than the primary diagnosis of cancer
* Weight < 5 kilograms
* Previous participation in CHP-810

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2004-06

PRIMARY OUTCOMES:
Characterization of Plasma Pharmacokinetics to examine the optimal dosing, metabolites and inter-patient variability of actinomycin-D in children with cancer during any sample of chemotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Abramson Research Center, Philadelphia, Pennsylvania, United States